CLINICAL TRIAL: NCT06757673
Title: Effectiveness of Robot-assisted Interaction Compared to Sensory Integration for Social Emotion Control in Autism Spectrum Disorder
Brief Title: Effectiveness of Robot-Assisted Intervention and Sensory Integration Therapy in Enhancing Social-Emotional Skills in Children With Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Yunlin University of Science and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202410030RINE
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Emotional Regulation; Sensory Integration Dysfunction
Keywords: Autism Spectrum Disorder; Sensory Integration; Robot-Assisted Therapy; Social-Emotional Skills; Early Intervention; Occupational Therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-Assisted Intervention (Experimental): Participants in this group will engage with the Kebbi Air smart robot, which delivers scripted social-emotional skill-building activities over a 12-week period.
  Interventions: Device: Robot-Assisted Therapy using Kebbi Air
- Sensory Integration Therapy (Active Comparator): Participants in this group will receive traditional sensory integration therapy, guided by occupational therapists, focusing on improving sensory processing and social-emotional regulation.
  Interventions: Behavioral: Sensory Integration Therapy

INTERVENTIONS:
Device: Robot-Assisted Therapy using Kebbi Air — Participants in this group will engage with the Kebbi Air smart robot, which is programmed with interactive scripts designed to enhance social-emotional regulation skills. The intervention includes weekly 30-minute sessions over a 12-week period, where the robot simulates real-life social scenarios and provides verbal and visual responses to guide participants in developing emotional and social skills. Occupational therapists will supervise these sessions to ensure the appropriateness of interactions and provide additional support as needed.
  Arms: Robot-Assisted Intervention
Behavioral: Sensory Integration Therapy — Participants in this group will receive traditional sensory integration therapy guided by occupational therapists. The therapy focuses on improving sensory processing and emotional regulation through structured activities targeting visual, auditory, and tactile stimuli. Each session is conducted weekly, lasting 30 minutes, for a total of 12 weeks. The therapy aims to help children adapt to sensory inputs and enhance their ability to engage in social interactions and manage emotions effectively.
  Arms: Sensory Integration Therapy

SUMMARY:
This study is designed to evaluate and compare the impact of robot-assisted intervention using a smart robot (Kebbi Air) and traditional sensory integration therapy on improving social-emotional skills in children diagnosed with autism spectrum disorder (ASD) or suspected ASD. The study will enroll children aged 4 to 6 years, who will be randomly assigned to one of two groups: the experimental group, which will participate in guided interactions with the smart robot, or the control group, which will receive sensory integration therapy tailored to enhance emotional and social functioning.

The research aims to explore whether interactions with the robot, which are designed to simulate real-world social scenarios, can provide comparable or enhanced benefits compared to traditional sensory integration methods. Pre- and post-intervention assessments will be conducted over a 12-week period, using tools like the Achenbach System of Empirically Based Assessment (ASEBA) and the Sensory Processing Measure (SPM) to measure changes in emotional regulation, sensory processing abilities, and social engagement. The study hypothesizes that the robot-assisted intervention will offer a novel, engaging, and effective approach to supporting the developmental needs of children with ASD.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of robot-assisted intervention compared to traditional sensory integration therapy in improving social-emotional regulation skills in children aged 4-6 years diagnosed with autism spectrum disorder (ASD) or suspected ASD. The research is designed as a randomized controlled trial with 12 participants divided into two groups: the experimental group and the control group.

Participants in the experimental group will interact with a smart robot (Kebbi Air) equipped with interactive scripts tailored to simulate real-life social scenarios. These interactions aim to teach emotional regulation and social skills through structured, engaging activities. The control group will receive sensory integration therapy provided by occupational therapists, focusing on enhancing sensory processing and emotional stability through activities targeting visual, auditory, and tactile stimuli.

The intervention will be conducted over a period of 12 weeks, with participants attending weekly 30-minute sessions. Assessments will be conducted before and after the intervention to measure its impact. Tools such as the Achenbach System of Empirically Based Assessment (ASEBA) and the Sensory Processing Measure (SPM) will be used to evaluate changes in emotional regulation, sensory processing, and social skills.

This study hypothesizes that the robot-assisted intervention will be as effective as or even superior to traditional sensory integration therapy, offering an engaging alternative for children with ASD. By combining cutting-edge technology with therapeutic strategies, the research seeks to provide insights into innovative approaches for supporting children's development, with the potential to inform future practices and interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-6 years, regardless of gender.
2. Diagnosed with autism spectrum disorder (ASD) or suspected ASD.
3. Cognitive ability: Developmental Quotient (DQ) ≥ 70, as assessed by the Comprehensive 4. Developmental Inventory for Infants and Toddlers (CDIIT).Social-emotional ability: DQ < 85, as assessed by CDIIT, indicating challenges in emotional regulation and social skills.

5. No significant physical or psychological conditions that could interfere with participation in the intervention.

Exclusion Criteria:

1. Children younger than 4 years or older than 6 years.
2. Cognitive ability: DQ < 70, as assessed by CDIIT, indicating limited learning potential.
3. Social-emotional ability: DQ ≥ 85, as assessed by CDIIT, indicating normal emotional and social functioning.
4. Any physical or psychological condition deemed by the investigators to interfere with the intervention or assessments.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Social-Emotional Regulation Skills | Baseline (pre-intervention) and after 12 weeks (post-intervention).
  Changes in emotional regulation, including anxiety, withdrawal, and aggression, were assessed using the Achenbach System of Empirically Based Assessment (ASEBA), specifically the Child Behavior Checklist for Ages 1½-5 (CBCL/1½-5). This caregiver-reported tool evaluates behavioral and emotional functioning in children aged 1.5 to 5 years. It assesses seven syndrome scales, including Emotional Reactivity, Anxiety/Depression, Somatic Complaints, Withdrawal, Attention Problems, Aggressive Behavior, and Sleep Problems. DSM-oriented scales identify issues such as affective, anxiety, and attention-deficit/hyperactivity problems. Items are rated on a 3-point Likert scale (0 = Not True, 1 = Somewhat True, 2 = Very True), with higher scores indicating greater severity. This tool tracks changes in emotional regulation over time.
Sensory Processing Abilities | Baseline (pre-intervention) and after 12 weeks (post-intervention).
  Sensory processing challenges and their impact on social participation were evaluated using the Sensory Processing Measure (SPM), a standardized tool for children aged 5 to 12 years. The SPM identifies sensory difficulties across domains: Social Participation, Vision, Hearing, Touch, Body Awareness (Proprioception), Balance and Motion (Vestibular), and Planning and Ideas (Praxis). Items are rated on a 4-point Likert scale (1 = Never, 4 = Always). Scores are categorized as Typical, Some Problems, or Definite Dysfunction, with higher scores indicating greater challenges. The SPM provides insights into how sensory processing affects a child's behavior and participation across various environments.

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet decided whether to share Individual Participant Data (IPD). The primary reasons include the need to consider privacy protection regulations, institutional policies, and the sensitive nature of the collected data. Additionally, the investigators need to ensure that data sharing can be conducted in compliance with ethical guidelines. The research team plans to evaluate the feasibility of data sharing after the study is completed, taking into account practical considerations and recommendations from regulatory authorities or ethics committees.